CLINICAL TRIAL: NCT01456793
Title: Evaluation of the Effectiveness of the Teen Options to Prevent Pregnancy (T.O.P.P.) Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mathematica Policy Research, Inc. (Other)
Collaborators: OhioHealth Research and Innovation Institute (Unknown); Nationwide Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MPR-06549-1
Record Dates: First submitted 2011-10-14; First posted 2011-10-21 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Pregnancy
Keywords: Pregnancy prevention; Pregnancy; Birth; Contraceptive use; Adolescents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Teen Options to Prevent Pregnancy (Experimental)
  Interventions: Behavioral: Teen Options to Prevent Pregnancy (T.O.P.P.)
- Usual care services (No Intervention)

INTERVENTIONS:
Behavioral: Teen Options to Prevent Pregnancy (T.O.P.P.) — Telephone-based care coordination and mobile contraceptive services
  Arms: Teen Options to Prevent Pregnancy

SUMMARY:
The purpose of this study is to evaluate the effectiveness of the Teen Options to Prevent Pregnancy (T.O.P.P.) program in increasing contraceptive use and reducing repeat pregnancies among pregnant and parenting adolescents in central Ohio.

DETAILED DESCRIPTION:
The risk for teen pregnancy is especially high among teen mothers, leading, in some cases, to unsafe intervals between teen births. The Teen Options to Prevent Pregnancy (T.O.P.P.) program is an 18-month clinic-based program that aims to reduce repeat pregnancies among pregnant and parenting adolescents by providing telephone-based care coordination and mobile contraceptive services to this high-risk population. This study uses a randomized controlled design to compare the effectiveness of T.O.P.P. versus usual care provided to patients at participating clinics. Study participants will be adolescent mothers between the ages of 10 to 19 recruited through seven OhioHealth women's health clinics and three OhioHealth hospitals covering seven counties in central Ohio. This study is being conducted as part of the national Evaluation of Adolescent Pregnancy Prevention Approaches funded by the U.S. Department of Health and Human Services' Office of Adolescent Health.

ELIGIBILITY:
Inclusion Criteria:

* 10 - 19 years old
* Female
* 28 weeks pregnant through 8 week post partum
* Medicaid recipient
* English speaking
* Patient of OhioHealth

Ages: 10 Years to 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 598 (Actual)
Dates: Start 2011-10; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Incidence of repeat pregnancy | 30 months after baseline

SECONDARY OUTCOMES:
Contraceptive Use | 6 months after baseline
Contraceptive Use | 18 months after baseline
Contraceptive Use | 30 months after baseline

CONTACTS AND LOCATIONS:
Overall Officials: Brian Goesling, PhD, Principal Investigator — Mathematica Policy Research; Jack Stevens, PhD, Principal Investigator — Nationwide Children's Hospital; Ngozi Osuagwu, MD, Principal Investigator — OhioHealth; Kimberly V Smith, PhD, Principal Investigator — Mathematica Policy Research
Locations (1):
- OhioHealth Community Partnerships, Columbus, Ohio, United States

REFERENCES:
- [Derived] Stevens J, Rotz D, Goesling B. Brief report: Assessing the risk of reporting bias in a RCT for adolescent mothers. J Adolesc. 2019 Jul;74:197-200. doi: 10.1016/j.adolescence.2019.06.011. Epub 2019 Jun 26. PMID 31252347
- [Derived] Stevens J, Lutz R, Osuagwu N, Rotz D, Goesling B. A randomized trial of motivational interviewing and facilitated contraceptive access to prevent rapid repeat pregnancy among adolescent mothers. Am J Obstet Gynecol. 2017 Oct;217(4):423.e1-423.e9. doi: 10.1016/j.ajog.2017.06.010. Epub 2017 Jun 12. PMID 28619692